CLINICAL TRIAL: NCT01882595
Title: Influence of Tracheostomy on Lung Deposition in Spontaneously Breathing Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, laurentpitance, Doctor in physiotherapy, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Nebu Tracheo
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Tracheostomized Patients
Keywords: Nebulization aerosol nebulizer tracheostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebulization through the tracheostomy (Experimental): Each subjects received two nebulization sessions. The first session was performed prior the tracheostomy removal (through the tracheostomy) and the second one when the when the tracheostome was totally scared (through the mouth)
  Interventions: Other: Nebulization through the tracheostomy
- Nebulization through the mouth (Active Comparator): Each subjects received two nebulization sessions. The first session was performed prior the tracheostomy removal (through the tracheostomy) and the second one when the when the tracheostome was totally scared (through the mouth)
  Interventions: Other: Nebulization through the mouth

INTERVENTIONS:
Other: Nebulization through the tracheostomy — Each subject received two nebulization sessions under spontaneous breathing in a sitting position. The first session was performed prior to tracheostomy removal. During the first nebulization, subjects inhaled the aerosol through the tracheostomy, cuff inflated and inner cannula removed.
  Arms: Nebulization through the tracheostomy
Other: Nebulization through the mouth — Each subject received two nebulization sessions under spontaneous breathing in a sitting position. The second nebulization was performed when the tracheostome was totally scarred. During the second nebulization, subjects inhaled the aerosol a mouth piece and wore a nose clip.
  Arms: Nebulization through the mouth

SUMMARY:
To compare lung deposition of amikacin in two settings: spontaneously breathing through a tracheostomy cannula and through the mouth.

ELIGIBILITY:
Inclusion Criteria:

* Patient who were likely to require an elective tracheostomy surgery as part as their head and neck surgery

Exclusion Criteria:

* Allergy to Aminoglycosides
* Patients who received Aminoglycosides treatment less than one month prior the surgery
* Pectoralis major flap reconstruction
* Latissimus dorsi flap reconstruction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-01; Primary Completion 2009-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Amikacin urinary drug concentration | At each micturition during 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium